CLINICAL TRIAL: NCT03530293
Title: A Phase 2, Double-Blind, Placebo-Controlled, Randomized Withdrawal Study to Evaluate the Safety and Efficacy of NBI-98854 in Pediatric Subjects With Tourette Syndrome
Brief Title: Safety and Efficacy of NBI-98854 in Pediatric Subjects With Tourette Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NBI-98854-TS2005
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: open-label study drug treatment period followed by blinded randomization into treatment arm or placebo arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pre-randomization Valbenazine (Experimental): Participants received valbenazine once daily for up to 12 weeks, depending on if and when randomization occured. The starting dose was 20 mg for participants <50 kg at baseline and 40 mg for participants ≥50 kg at baseline, and could be escalated in increments of 20 mg every 2 weeks to a maximum of 60 mg for participants <50 kg and 80 mg for participants ≥50 kg to achieve an optimal dose of valbenazine for each participant.
  Interventions: Drug: Valbenazine
- Randomized Placebo (Placebo Comparator): Participants received placebo (matching valbenazine) once daily from randomization (Week 8, 10, or 12) through Week 36. Randomization into this arm occurred after treatment with valbenazine once daily through randomization.
  Interventions: Drug: Placebo oral capsule
- Randomized Valbenazine (Experimental): Participants received their optimized dose of valbenazine once daily from randomization (Week 8, 10, or 12) through Week 36. Randomization into this arm occurred after treatment with valbenazine once daily through randomization.
  Interventions: Drug: Valbenazine

INTERVENTIONS:
Drug: Valbenazine — vesicular monoamine transporter 2 (VMAT2) inhibitor
  Other Names: NBI-98854
  Arms: Pre-randomization Valbenazine; Randomized Valbenazine
Drug: Placebo oral capsule — non-active dosage form
  Arms: Randomized Placebo

SUMMARY:
This is a Phase 2, double-blind, placebo-controlled, randomized withdrawal study to evaluate the safety and maintenance of efficacy of an optimized once-daily (qd) dose of NBI-98854 in pediatric subjects with TS.

ELIGIBILITY:
Inclusion Criteria:

1. Have a clinical diagnosis of Tourette Syndrome (TS)
2. Have at least moderate tic severity
3. Have TS symptoms that impair school, occupational, and/or social function
4. If using maintenance medication(s) for TS or TS spectrum diagnoses (e.g. obsessive-compulsive disorder [OCD], Attention-Deficit Hyperactivity Disorder [ADHD]), be on stable doses
5. Be in good general health
6. Adolescent subjects (12 to 17 years of age) must have a negative urine drug screen for amphetamines, barbiturates, benzodiazepine, phencyclidine, cocaine, opiates, or cannabinoids and a negative alcohol screen
7. Subjects of childbearing potential who do not practice total abstinence must agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently during the screening, treatment and follow-up periods of the study

Exclusion Criteria:

1. Have an active, clinically significant unstable medical condition within 1 month prior to screening
2. Have a known history of long QT syndrome or cardiac arrhythmia
3. Have a known history of neuroleptic malignant syndrome
4. Have a cancer diagnosis within 3 years prior to screening (some exceptions allowed)
5. Have an allergy, hypersensitivity, or intolerance to VMAT2 inhibitors
6. Have a blood loss ≥250 mL or donated blood within 30 days prior to screening
7. Have a known history of substance dependence, substance (drug) or alcohol abuse
8. Have a significant risk of suicidal or violent behavior
9. Have initiated Comprehensive Behavioral Intervention for Tics (CBIT) during the screening period or at baseline or plan to initiate CBIT during the study
10. Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than NBI-98854) during the study
11. Have previously participated in an NBI-98854 clinical study, except for NBI-98854-1403 or NBI-98854-1501.
12. Have HIV, hepatitis B, or hepatitis C

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (47):
- United States (46):
  - Neuricrine Clinical Site, Sun City, Arizona
  - Neurocrine Clinical Site, Little Rock, Arkansas
  - Neurocrine Clinical Site, Rogers, Arkansas
  - Neurocrine Clinical Site, Anaheim, California
  - Neurocrine Clinical Site, Fullerton, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, Santa Ana, California
  - Neurocrine Clinical Site, Pueblo, Colorado
  - Neurocrine Clinical Site, Stamford, Connecticut
  - Neurocrine Clinical Site, Washington D.C., District of Columbia
  - Neurocrine Clinical Site, Gulf Breeze, Florida
  - Neurocrine Clinical Site, Hialeah, Florida
  - Neurocrine Clinical Site, Miami, Florida
  - Neurocrine Clinical Site, North Miami, Florida
  - Neurocrine Clinical Site, Orlando, Florida
  - Neurocrine Clinical Site, Palmetto Bay, Florida
  - Neurocrine Clinical Site, Spring Hill, Florida
  - Neurocrine Clinical Site, St. Petersburg, Florida
  - Neurocrine Clinical Site, Tallahassee, Florida
  - Neurocrine Clinical Site, Atlanta, Georgia
  - Neurocrine Clinical Site, Fayetteville, Georgia
  - Neurocrine Clinical Site, Savannah, Georgia
  - Neurocrine Clinical Site, Chicago, Illinois
  - Neurocrine Clinical Site, South Bend, Indiana
  - Neurocrine Clinical Site, Boston, Massachusetts
  - Neurocrine Clinical Site, Ann Arbor, Michigan
  - Neurocrine Clinical Site, Bloomfield Hills, Michigan
  - Neurocrine Clinical Site, West Bloomfield, Michigan
  - Neurocrine Clinical Site, Lincoln, Nebraska
  - Neurocrine Clinical Site, Nashua, New Hampshire
  - Neurocrine Clinical Site, Cherry Hill, New Jersey
  - Neurocrine Clinical Site, Mount Arlington, New Jersey
  - Neurocrine Clinical Site, New York, New York
  - Neurocrine Clinical Site, South Setauket, New York
  - Neurocrine Clinical Site, Charlotte, North Carolina
  - Neurocrine Clinical Site, Mason, Ohio
  - Neurocrine Clinical Site, Oklahoma City, Oklahoma
  - Neurocrine Clinical Site, Dallas, Texas
  - Neurocrine Clinical Site, DeSoto, Texas
  - Neurocrine Clinical Site, Houston, Texas
  - Neurocrine Clinical Site, Irving, Texas
  - Neurocrine Clinical Site, San Antonio, Texas
  - Neurocrine Clinical Site, Charlottesville, Virginia
  - Neurocrine Clinical Site, Bothell, Washington
  - Neurocrine Clinical Site, Everett, Washington
  - Neurocrine Clinical Site, Spokane, Washington
- Neurocrine Clinical Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 180 male and female pediatric subjects between 6 and 17 years of age (inclusive) with a DSM-IV or -V diagnosis of TS were planned to be enrolled. A total of 81 subjects were enrolled. The first and last participants were enrolled on April 17 2018 and May 7 2019, respectively.
Pre-assignment Details: At the end of Weeks 8, 10, or 12, treatment responders (sufficient control of tic behaviors based on investigator assessment) were randomized in a 1:1 ratio to placebo or valbenazine. Randomization was stratified based on the subject's weight group at baseline (<50 kg versus ≥50 kg). The visit week when subjects were randomized was blinded. At Week 12 all nonresponders were discontinued.
Groups:
- Pre-randomization Valbenazine: Participants received valbenazine once daily for up to 12 weeks, depending on if and when randomization occurred. The starting dose was 20 mg for participants <50 kg at baseline and 40 mg for participants ≥50 kg at baseline, and could be escalated in increments of 20 mg every 2 weeks to a maximum of 60 mg for participants <50 kg and 80 mg for participants ≥50 kg to achieve an optimal dose of valbenazine for each participant.
Period: Pre-randomization
Arm/Group | Pre-randomization Valbenazine | Randomized Placebo | Randomized Valbenazine
Started | 81 | 0 | 0
Safety Analysis Set (The safety analysis set includes all enrolled subjects who received at least one dose of study drug and had any safety data collected after the first dose of study drug.) | 80 | 0 | 0
Completed | 57 | 0 | 0
Not Completed | 24 | 0 | 0
Not completed — Adverse Event | 12 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Study Terminated by Sponsor | 5 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0
Period: Randomized Withdrawal Period / Follow-up
Arm/Group | Pre-randomization Valbenazine | Randomized Placebo | Randomized Valbenazine
Started (5 subjects completed the pre-randomization period but were ineligible for randomization due to lack of response.) | 0 | 26 | 26
Completed | 0 | 9 | 9
Not Completed | 0 | 17 | 17
Not completed — Adverse Event | 0 | 2 | 4
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 2
Not completed — Lack of Efficacy | 0 | 2 | 0
Not completed — Study Terminated by Sponsor | 0 | 10 | 10

BASELINE CHARACTERISTICS:
Population: The full analysis set includes all subjects who were randomized to a treatment group and had at least one post-randomization visit where loss of treatment response was able to be assessed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Placebo | Randomized Valbenazine | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.7 (2.7) | 12.8 (3.1) | 12.8 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 21 | 24 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 22 | 24 | 46
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Loss of Treatment Response
Description: Loss of treatment response during the withdrawal period was defined as: 2 consecutive visits with 1) an increase in the Yale Global Tic Severity Scale (YGTSS) Total Tic Score (TTS) of greater than 35% or 7 points from the randomized withdrawal period baseline and 2) an increase in CGI-Tics-Severity score of ≥2 points from the randomized withdrawal period baseline; or discontinuation due to lack of efficacy or a treatment-emergent adverse event (TEAE) of worsening of tics. Median (lower and upper quartiles) Kaplan-Meier estimates for the time to loss of treatment response were not able to be calculated because of the low incidence of loss of treatment response events.
Time Frame: Randomization (Week 8, 10 or 12) through Week 36
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Randomized Placebo | Randomized Valbenazine
Number analyzed (Participants) | 26 | 26
Days | NA [NA to NA] — Kaplan-Meier estimates for the time to loss of treatment response were not able to be calculated because of the low incidence of loss of treatment response events. | NA [NA to NA] — Kaplan-Meier estimates for the time to loss of treatment response were not able to be calculated because of the low incidence of loss of treatment response events.

2. Secondary Outcome: Change From Randomization Baseline to the 8 Weeks Post-randomization Timepoint in the YGTSS TTS
Description: The YGTSS is designed to rate the overall severity of motor and phonic tic symptoms across a range of dimensions: number, frequency, intensity, complexity, and interference. The YGTSS was administered by the investigator (or qualified designee) using a computer-based structured clinical interview. The TTS is the sum of the 5 motor tic items and the 5 phonic (vocal) tic items and ranges from 0 to 50, with higher scores representing greater severity. Least-squares mean were estimated using a mixed-effects model for repeated measures.
Time Frame: Randomization Baseline (Week 8, 10 or 12); 8 weeks post-randomization
Population: The full analysis set includes all subjects who were randomized to a treatment group and had at least one post-randomization visit where loss of treatment response was able to be assessed. Participants who do not have a TTS value at a scheduled or mapped early termination visit after randomization are not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Randomized Placebo | Randomized Valbenazine
Number analyzed (Participants) | 26 | 25
units on a scale | 3.8 (1.6) | -1.0 (1.7)

3. Secondary Outcome: Change From Randomization Baseline to the Week 36 Visit in the YGTSS TTS
Description: The YGTSS is designed to rate the overall severity of motor and phonic tic symptoms across a range of dimensions: number, frequency, intensity, complexity, and interference. The YGTSS was administered by the investigator (or qualified designee) using a computer-based structured clinical interview. The TTS is the sum of the 5 motor tic items and the 5 phonic (vocal) tic items and ranges from 0 to 50, with higher scores representing greater severity.
Time Frame: Randomization Baseline (Week 8, 10 or 12); Week 36
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Placebo | Randomized Valbenazine
Number analyzed (Participants) | 9 | 9
units on a scale | 0.6 (12.06) | 0.1 (8.21)

4. Secondary Outcome: Change From Randomization Baseline to the 8 Weeks Post-randomization Timepoint in the CGI-Tics-Severity Score
Description: The CGI-Tics-Severity scale is used to assess overall severity on a 7-point scale. Each of the CGI-Tics-Severity response categories was assigned a numerical score as follows: 1 = Normal, not at all ill; 2 = Borderline ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; 7 = Among the most extremely ill patient.
Time Frame: Randomization Baseline (Week 8, 10 or 12); 8 weeks post-randomization
Population: The full analysis set includes all subjects who were randomized to a treatment group and had at least one post-randomization visit where loss of treatment response was able to be assessed. Participants who do not have a CGI-Tics-Severity value at a scheduled or mapped early termination visit after randomization are not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Randomized Placebo | Randomized Valbenazine
Number analyzed (Participants) | 22 | 19
units on a scale | 0.7 (0.2) | -0.1 (0.2)

5. Secondary Outcome: Change From Randomization Baseline to the Week 36 Visit in the CGI-Tics-Severity Score
Description: as for outcome 4
Time Frame: Randomization Baseline (Week 8, 10 or 12); Week 36
Population: The full analysis set includes all subjects who were randomized to a treatment group and hac at least one post-randomization visit where loss of treatment response was able to be assessed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Placebo | Randomized Valbenazine
Number analyzed (Participants) | 9 | 9
units on a scale | 0.1 (0.78) | 0.2 (1.30)

ADVERSE EVENTS:
Time Frame: Pre-randomization valbenazine group: from baseline up to randomization (Week 8, 10 or 12) or end of participation in subjects who did not randomize, up to 16 weeks. Randomized placebo and valbenazine groups: from randomization (Week 8, 10 or 12) up to Week 40
Groups:
- Pre-randomization Valbenazine: Participants received valbenazine once daily for up to 12 weeks, depending on if and when randomization occurs. The starting dose was 20 mg for participants <50 kg at baseline and 40 mg for participants ≥50 kg at baseline, and could be escalated in increments of 20 mg every 2 weeks to a maximum of 60 mg for subjects <50 kg and 80 mg for subjects ≥50 kg to achieve an optimal dose of valbenazine for each participant.
  Valbenazine: vesicular monoamine transporter 2 (VMAT2) inhibitor
Arm/Group | Pre-randomization Valbenazine | Randomized Placebo | Randomized Valbenazine
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/80 | 2/26 | 2/26
Other Adverse Events (participants affected / at risk) | 41/80 | 12/26 | 14/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-randomization Valbenazine (N=80) | Randomized Placebo (N=26) | Randomized Valbenazine (N=26)
Enterovirus infection (Infections and infestations) | 1 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 1
Tic (Psychiatric disorders) | 0 | 0 | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 1 | 0
Tourette's disorder (Congenital, familial and genetic disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-randomization Valbenazine (N=80) | Randomized Placebo (N=26) | Randomized Valbenazine (N=26)
Nausea (Gastrointestinal disorders) | 4 | 1 | 4
Vomiting (Gastrointestinal disorders) | 4 | 0 | 3
Fatigue (General disorders) | 10 | 1 | 0
Irritability (General disorders) | 6 | 4 | 4
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2
Weight increased (Investigations) | 6 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Headache (Nervous system disorders) | 9 | 3 | 2
Somnolence (Nervous system disorders) | 20 | 0 | 1
Aggression (Psychiatric disorders) | 1 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 4 | 0
Insomnia (Psychiatric disorders) | 5 | 2 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 2
Tic (Psychiatric disorders) | 1 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT03530293/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT03530293/SAP_001.pdf